CLINICAL TRIAL: NCT05429814
Title: Topical Menthol Application in Chemotherapy-Related Peripheral Neuropathy in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Deniz Ozdemir, Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21129002
Record Dates: First submitted 2022-06-11; First posted 2022-06-23 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Peripheral Neuropathies; Chemotherapy Effect
Keywords: Breast Cancer; Peripheral neuropathy; Menthol; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): During the study, the patients' routine pharmacological treatments will continue and menthol will be applied only to reduce the effect of neuropathy. In the study, menthol 1% will be used topically, as it was used in studies after the literature review. Although it was stated in the studies that menthol had no side effects, it was decided to mix menthol with water-based cream according to the literature recommendation. Researchers will first determine how many grams of menthol will be sufficient by applying menthol to their hands and feet.After the gram of the prepared mixture is determined, it will be given to the patients. Patients in the intervention group will be taught how to regularly apply menthol cream (topical menthol) to their hands and feet, twice a day, every day. The effect on CIPN will be evaluated in patients with CIPN for 3 weeks immediately before and after 6 weeks of treatment with menthol administration.
  Interventions: Other: Menthol Application
- control group (No Intervention): control group will receive standard practice

INTERVENTIONS:
Other: Menthol Application — During the study, the patients' routine pharmacological treatments will continue and menthol will be applied only to reduce the effect of neuropathy. In the study, menthol 1% will be used topically, as it was used in studies after the literature review. Although it was stated in the studies that menthol had no side effects, it was decided to mix menthol with water-based cream according to the literature recommendation. Researchers will first determine how many grams of menthol will be sufficient by applying menthol to their hands and feet.After the gram of the prepared mixture is determined, it will be given to the patients. Patients in the intervention group will be taught how to regularly apply menthol cream (topical menthol) to their hands and feet, twice a day, every day. The effect on CIPN will be evaluated in patients with CIPN for 3 weeks immediately before and after 6 weeks of treatment with menthol administration.
  Arms: Experimental

SUMMARY:
Peripheral neuropathy resulting from chemotherapy is a problem that concerns not only the individual but also their relatives and all healthcare personnel responsible for care. Studies to be carried out in this area are important in terms of providing evidence for nurses' practices and supporting the individual by alleviating the symptoms of the disease. Based on this information, the aim of this study is to determine the effect of menthol application, which will be applied to the hands and feet of breast cancer patients receiving chemotherapy, on CIPN.

DETAILED DESCRIPTION:
Introduction and Aim: Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most common side effects of chemotherapeutic agents. CIPN is a frequently dose-limiting neurotoxicity that causes significant deterioration in patients' quality of life. CIPN mainly plays a role in sensory peripheral neuropathy, although some patients have motor symptoms such as weakness and autonomic neuropathy. Sensory neuropathy is often distributed in the form of socks and gloves, causing symptoms such as spontaneous pain, allodynia, hyperalgesia, hypoesthesia, pins and needles, numbness, paresthesia, tingling, and gait disturbance. Treatment of CIPN requires non-toxic therapies as most of the pharmacological treatments for neuropathic pain, including antidepressants and anticonvulsants, have toxic side effects. Patients seek supportive strategies in the management of CIPN. There are a limited number of studies on non-pharmacological methods such as cryotherapy, massage, acupuncture, henna on hands and feet used in the management of peripheral neuropathy. Menthol has been widely used in traditional medicine as a topical pain reliever since ancient times. Creams containing menthol are available in the form of liquid, gel or lotion. Menthol-containing products that have not been studied in CIPN management are used in patients with a wide variety of ailments, including muscle pain, back, joint pain, and management of arthritis-related pain. Recent advances in the pathophysiology of pain have revealed new pathways responsible for the analgesic effect of menthol. Therefore, it is very important to determine the basic science and clinical efficacy data on the pain-relieving and cooling properties of menthol. Menthol (mint camphor) is an essential oil extract obtained from the genus Mentha (mint). Oncology clinical practice guidelines (ESMO; EONS; EANO) used for the diagnosis, prevention, treatment and follow-up of peripheral neurotoxicity caused by systemic anticancer therapy recommend menthol as a local intervention. Although these guidelines recommend menthol application, no studies have been found in the national and international literature showing the effect of topical menthol application in chemotherapy-induced peripheral neuropathy in patients with breast cancer. Peripheral neuropathy resulting from chemotherapy is a problem that concerns not only the individual but also their relatives and all healthcare personnel responsible for care. Studies to be carried out in this area are important in terms of providing evidence for nurses' practices and supporting the individual by alleviating the symptoms of the disease. Based on this information, the aim of this study is to determine the effect of menthol application on CIPN, which will be applied to the hands and feet of breast cancer patients receiving chemotherapy.

Method: The project was planned as a prospective, single-blind, randomized controlled experimental type.

The research will be carried out in Konya Necmettin Erbakan University Meram Medical Faculty Hospital Oncology Department between November 2021 and November 2022. In determining the sample size, based on the studies in the literature, the minimum number of samples was determined as 60, 30 in each group, with 95% confidence, 80% test power, and considering possible losses. Questionnaire Form, Chemotherapy-Induced Peripheral Neuropathy Evaluation Tool (CIPNAT) will be used as data collection tools.

Management: Data will be collected by the assistant researcher at the beginning of the study, at 3 weeks and at 6 weeks, in the doctor's room in the Oncology building of Necmettin Erbakan University Meram Medical Faculty Hospital. In the preliminary application of the study, a questionnaire will be applied to 10 patients.

Menthol Application During the study, the patients' routine pharmacological treatments will continue and menthol will be applied only to reduce the effect of neuropathy. In the study, menthol 1% will be used topically, as it was used in studies after the literature review. Although it was stated in the studies that menthol had no side effects, it was decided to mix menthol with water-based cream according to the literature recommendation. Researchers will first determine how many grams of menthol will be sufficient by applying menthol to their hands and feet.After the gram of the prepared mixture is determined, it will be given to the patients. Patients in the intervention group will be taught how to regularly apply menthol cream (topical menthol) to their hands and feet, twice a day, every day. The effect on CIPN will be evaluated in patients with CIPN for 3 weeks immediately before and after 6 weeks of treatment with menthol administration.

Widespread effect: Studies have shown that topical menthol application reduces chemotherapy-induced peripheral neuropathy. It has been determined that 1% menthol cream, which is applied to the hands and feet twice a day, reduces the severity of neuropathy symptoms and reduces neuropathy pain. This study will contribute to the literature and will have a significant impact on the quality of life of many cancer patients and cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received at least two cycles of chemotherapy
* Patients aged 18 and over
* Women who received the paclitaxel chemotherapy protocol will be included.

Exclusion Criteria:

* Those with open wounds and edema on their hands and feet
* Patients with diabetes mellitus and peripheral neuropathy due to autoimmune disease
* Use complementary and alternative treatment methods to prevent peripheral neuropathy throughout the treatment process.
* Those who are allergic to topical menthol to be used in the study will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) | 3 weeks after the first assessment
  The first section assesses the nine main symptoms as well as their severity, the extent to which they cause emotional disruption, and the frequency of their occurrence. The first six items in this section are related to sensory symptoms, while the seventh, eighth and ninth items are related to sub-dimensions of motor symptoms. In the second part, 14 activities were evaluated and questions were asked about the effect level of these substances. The activities assessed included fine motor and general activities. To assess the symptoms listed in the first section, "Yes" was considered equal to 1 point and "No" equal to 0 (0-9); their severity, symptoms, extent and frequency of emotional impairment were scored between 0 and 10 (0-270). The total score for the first part of the instrument is between 0 and 279. The effect level on the 14 activities in the second part was calculated between 0 and 10 (0-140). The Cronbach's alpha value of the original scale is 0.95
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) | 6 weeks after the first assessment
  The first section assesses the nine main symptoms as well as their severity, the extent to which they cause emotional disruption, and the frequency of their occurrence. The first six items in this section are related to sensory symptoms, while the seventh, eighth and ninth items are related to sub-dimensions of motor symptoms. In the second part, 14 activities were evaluated and questions were asked about the effect level of these substances. The activities assessed included fine motor and general activities. To assess the symptoms listed in the first section, "Yes" was considered equal to 1 point and "No" equal to 0 (0-9); their severity, symptoms, extent and frequency of emotional impairment were scored between 0 and 10 (0-270). The total score for the first part of the instrument is between 0 and 279. The effect level on the 14 activities in the second part was calculated between 0 and 10 (0-140). The Cronbach's alpha value of the original scale is 0.95

CONTACTS AND LOCATIONS:
Overall Officials: Selda Arslan, Phd, Study Director — Necmettin Erbakan University Faculty of Nursing
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir D, Arslan S, Artac M, Karaarslan F. Topical menthol for chemotherapy-induced peripheral neuropathy: a randomised controlled trial in breast cancer. BMJ Support Palliat Care. 2024 Dec 25;15(1):79-86. doi: 10.1136/spcare-2023-004483. PMID 39038990